CLINICAL TRIAL: NCT01175668
Title: Comparison of Clonidine Versus Phenobarbital as an Adjunct Therapy for Neonatal Abstinence Syndrome
Brief Title: Clonidine for Neonatal Abstinence Syndrome Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Based on the planned interim analysis results at 50% recruitment, after IRB reviewed the results, further enrollment was stopped.
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Rachana Singh, MD, Assistant Professor of Pediatrics, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH-10-196
Record Dates: First submitted 2010-07-14; First posted 2010-08-05 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2013-11

CONDITIONS: Neonatal Abstinence Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Clonidine; Phenobarbital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NMS/Clonidine (Experimental)
  Interventions: Drug: Clonidine
- NMS/Phenobarbital (Active Comparator)
  Interventions: Drug: Phenobarbital

INTERVENTIONS:
Drug: Clonidine — This group of infants undergoing NAS will be treated with neonatal morphine sulfate and Clonidine as an adjunct medication to control the symptoms. Once stable Finnegan scores <8 for 24h, NMS will be weaned by 10% daily till off, then Clonidine will be weaned off in a stepwise manner. Infant will not go home on any medication for NAS. NMS will be dosed as mg/kd/day divided q3h and Clonidine will be dosed as microgm/kg/day divided q6h based upon the initial Finnegan scores.
  Arms: NMS/Clonidine
Drug: Phenobarbital — Infants in this arm will be treated as current standard practice with NMS and Phenobarbital. NMS will be weaned by 10% daily to completely off during the hospital stay. Infants will be discharged home on Phenobarbital.
  NMS will be dosed as mg/kg/day divided q3h and Phenobarbital will be dosed as mg/kg/day divided q8h based on the Finnegan scores.
  Arms: NMS/Phenobarbital

SUMMARY:
The study plans to compare the use of Clonidine versus Phenobarbital as an additional medication to neonatal morphine sulfate for treatment of newborn infants undergoing drug withdrawal symptoms due to mother's use of opioid drug use. The investigators hypothesis is that use of Clonidine will lead to shorter duration of treatment, hospital stay and thereby early discharge home.

DETAILED DESCRIPTION:
Introduction: Neonatal abstinence syndrome (NAS) is a symptom complex experienced by 55 to 94% of neonates who are exposed to intrauterine opioids. Recent studies have shown that combination therapies are superior to monotherapy with neonatal morphine sulfate (NMS). Phenobarbital has been shown to reduce the length of hospitalization, decrease severity of withdrawal, as well as decrease hospital costs and care giver demands. Similarly, clonidine, an α2-adrenergic receptor agonist, has also been shown to be safe, effective and reduces length of treatment.

Phenobarbital as an antiepileptic acts on the GABA (A) receptors and has been shown in animal models to inhibit neuronal cell proliferation, survival and neurogenesis. In human infants long term treatment with phenobarbital may result in neuro-developmental compromise. Due to these potentially harmful effects of Phenobarbital (P) alternative therapies should be explored more thoroughly including clonidine (C).

Our primary aim is to compare the length of NAS treatment with NMS in the two study groups - NMS/C versus NMS/P. Our secondary aims are to compare the total dosage of NMS, total length of hospital stay for NAS treatment, treatment failures and adverse effect profiles for the two study groups. We hypothesize that clonidine when compared to phenobarbital as an adjunct therapy, will have shorter length of stay, with fewer treatment failures and side effects.

Study design/Methods: This study will be a prospective, randomized, non-blinded clinical trial of NMS/C versus NMS/P for treatment of infants with NAS. Infants will be recruited from the Baystate Children's Hospital Neonatal Intensive Care Unit (NICU) and Neonatal Continuing Care Nursery (NCCN), a level III unit, over a 2 year study period. After randomization, infants will adhere to strict treatment initiation and withdrawal protocols. Maternal and infant descriptive data will be collected along with specific data regarding vital signs, drug dosages, length of treatment, treatment failures and adverse effects.

The primary outcome will be length of treatment with NMS in the two study arms. The secondary outcomes will be - a) total length of hospital stay for NAS treatment, b) mean total treatment dose and mean daily dose of NMS, c) total number of treatment failures,d) adverse effects such as bradycardia, hypotension, hypertension e) Total outpatient therapy days with Phenobarbital

Significance: This comparison study is potentially of great significance. If clonidine is proven to be equally effective in treatment of NAS many of the detrimental effects of phenobarbital therapy may be avoided for infants on long term pharmacotherapy for treatment of withdrawal with shorter length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 15 days of age
* Prenatal exposure to opioids with development of moderate to severe NAS (2 consecutive abstinence scores of ≥ 8)
* Medically stable

Exclusion Criteria:

* Gestational age < 35 weeks
* Intrauterine growth retardation (birth weight below the 5th percentile)
* Congenital heart disease
* Congenital anomalies
* Medically unstable

Exposure to Benzodiazepines prenatally

-

Max Age: 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2010-07; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachana Singh, MD, MS, Principal Investigator — Baystate Medical Center
Locations (1):
- NICU @ Baystate Children's Hospital, Springfield, Massachusetts, United States

REFERENCES:
- [Result] Surran B, Visintainer P, Chamberlain S, Kopcza K, Shah B, Singh R. Efficacy of clonidine versus phenobarbital in reducing neonatal morphine sulfate therapy days for neonatal abstinence syndrome. A prospective randomized clinical trial. J Perinatol. 2013 Dec;33(12):954-9. doi: 10.1038/jp.2013.95. Epub 2013 Aug 15. PMID 23949834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at Baystate Children's Hospital Davis Neonatal Intensive Care Unit (NICU), a level III, regional perinatal referral center, for Western Massachusetts, from June 2010 to June 2012
Pre-assignment Details: Overall 82 infants were consented for the study but 14 were excluded either because they did not have continued high modified Finnegan Scores (n=13), or had Unstable clinical status (n=1)
Groups:
- NMS/Clonidine: Dosing was based on the Finnegan scores as below
  Finn Score 8-10 NMS 0.32mg/kg/day + Clonidine 6 mcg/kg/day 11-13 NMS 0.48 mg/kg/day + Clonidine 8 mcg/kg/day 14-16 NMS 0.64 mg/kg/day + Clonidine 10 mcg/kg/day ≥17 NMS 0.8 mg/kg/day* + Clonidine 12 mcg/kg/day
  Daily NMS dose was divided for q3h dosing interval Daily Clonidine dose was divided for q6h dosing interval Clonidine escalation may be limited by hypotension or bradycardia
  *If needing morphine sulfate > 0.8 mg/kg/day, increase dose in increments of 0.16 mg/kg/day until Finnegan score < 8
- NMS/Phenobarbital: Dosing was based on the Finnegan scores as below
  Finn Score 8-10 NMS 0.32mg/kg/day +Phenobarbital 6 mg/kg/day 11-13 NMS 0.48 mg/kg/day +Phenobarbital 8 mg/kg/day 14-16 NMS 0.64 mg/kg/day +Phenobarbital 10 mg/kg/day ≥17 NMS 0.8 mg/kg/day* + Phenobarbital 12 mg/kg/day
  Daily NMS dose was divided for q3h dosing interval Daily Phenobarbital dose was divided for q8h dosing interval
  *If needing morphine sulfate > 0.8 mg/kg/day, increase dose in increments of 0.16 mg/kg/day until Finnegan score < 8
Period: Overall Study
Arm/Group | NMS/Clonidine | NMS/Phenobarbital
Started | 34 | 34
Completed | 32 | 34
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NMS/Clonidine | NMS/Phenobarbital | Total
Number analyzed (Participants) | 34 | 34 | 68
Age Continuous [Mean (Standard Deviation); unit: days] | 1.8 (0.9) | 2.26 (1.60) | 2.05 (1.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Length of Treatment With Neonatal Morphine Sulfate
Time Frame: subjects were followed for the duration of treatment, up to 3 months
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | NMS/Clonidine | NMS/Phenobarbital
Number analyzed (Participants) | 32 | 34
days | 18.2 [14.9 to 21.5] | 13.6 [11.0 to 16.1]

2. Secondary Outcome: Total Dose of NMS Used
Time Frame: For the duration of treatment, upto 3 months
Measure: Mean (95% Confidence Interval); unit: mg/kg
Arm/Group | NMS/Clonidine | NMS/Phenobarbital
Number analyzed (Participants) | 32 | 34
mg/kg | 5.7 [4.7 to 6.8] | 4.6 [3.8 to 5.4]

ADVERSE EVENTS:
Time Frame: During the hospital stay
Description: In the phenobarbital group, 3 infants (8.8%), manifested over sedation signs (poor feeds, and mild respiratory depression). This prompted serum phenobarbital measurements which were noted to be supra-therapeutic (>40 mg/dL) and required dosage adjustment.
Arm/Group | NMS/Clonidine | NMS/Phenobarbital
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 3/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NMS/Clonidine (N=34) | NMS/Phenobarbital (N=34)
Oversedation (Nervous system disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
One of the major limitations to our study was the inability to blind the two groups for the study medications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No